CLINICAL TRIAL: NCT01996761
Title: Effects of Cerebrolysin on Motor Recovery in Patients With Subacute Stroke
Acronym: E-COMPASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Yun-Hee Kim, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-09-084-001
Record Dates: First submitted 2013-11-05; First posted 2013-11-27 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Cerebrolysin
MeSH Terms: interventions — cerebrolysin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Study Group 1 (Experimental): Study Group 1: 30ml Cerebrolysin
  Interventions: Drug: porcine brain peptide (Cerebrolysin)
- Study Group 2 (Placebo Comparator): Study Group 2: Placebo (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: porcine brain peptide (Cerebrolysin)
  Arms: Study Group 1
Drug: Placebo
  Arms: Study Group 2

SUMMARY:
This study, E-COMPASS is a phase IV clinical trial designed as a multicenter, randomized, double-blind, placebo-controlled, parallel-group study. This study will enroll 75 subacute stroke patients with unilateral motor dysfunction. Primary objective is to demonstrate the efficacy of porcine brain peptide to improve motor recovery measured by the improvement ratio of Fugl-Meyer assessment ((score of FMA after 3 weeks - score of FMA at baseline) / score of FMA at baseline) in patients with subacute stroke.

ELIGIBILITY:
Inclusion Criteria:

1. 1st cortical or subcortical unilateral infarction (supratentorial lesion)
2. Confirmed by CT or MRI
3. Subacute stage: less than 1 week
4. Moderate to severe motor function involvement-total of FMA: 0-84
5. Age: between 18 and 80 years
6. Inpatients

Exclusion Criteria:

1. Progressive or unstable stroke
2. Pre-existing and active major neurological disease
3. Pre-existing and active (e.g., on chronic medication) major psychiatric disease, such as major depression, schizophrenia, bipolar disease, or dementia
4. A history of significant alcohol or drug abuse in the prior 3 years
5. Advanced liver, kidney, cardiac, or pulmonary disease
6. A terminal medical diagnosis consistent with survival < 1 year
7. Substantial decrease in alertness at the time of randomization, defined as score of 2 on NIH Stroke Scale
8. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female in reproductive years
9. Any condition that would represent a contraindication to Cerebrolysin, including allergy to Cerebrolysin
10. Current enrolment in another therapeutic study of stroke or stroke recovery
11. Total serum bilirubin > 4 mg/dL, alkaline phosphatase > 250 U/L, SGOT/AST > 150 U/L, SGPT/ALT > 150 U/L, or creatinine > 3.5 mg/dL; or cardiopulmonary deficits large enough to interfere with reasonable participation in physiotherapy during the trial.
12. Previous porcine brain peptide administration history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
the improvement ratio of Fugl-Meyer assessment | after 3 weeks
  Primary objective is to demonstrate the efficacy of porcine brain peptide to improve motor recovery measured by the improvement ratio of Fugl-Meyer assessment ((score of FMA after 3 weeks - score of FMA at baseline) / score of FMA at baseline) in patients with subacute stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Chang WH, Park CH, Kim DY, Shin YI, Ko MH, Lee A, Jang SY, Kim YH. Cerebrolysin combined with rehabilitation promotes motor recovery in patients with severe motor impairment after stroke. BMC Neurol. 2016 Mar 2;16:31. doi: 10.1186/s12883-016-0553-z. PMID 26934986